CLINICAL TRIAL: NCT06024538
Title: Role of Cancer-associated Fibroblast, MDSCs and Immune Cell Interplays in the Resistance of Non-small Cell Lung Cancer to Anti-PD1/PD-L1 Therapies
Acronym: COCKPI-T
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/34
Record Dates: First submitted 2023-08-28; First posted 2023-09-06 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Lung Neoplasm; Cancer Associated Fibroblast; Myeloid-Derived Suppressive Cells Immunosuppression
Keywords: Lung cancer; Immunosuppression; Immunotherapy; Immuno-oncology; Antitumor immune escape
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective part of the study
  Interventions: Procedure: Tumor samples

INTERVENTIONS:
Procedure: Tumor samples — Tumor samples will be collected by the pathologist at the reception of the tumor removed during surgery

SUMMARY:
Immunotherapy have revolutionized the field of oncology, but response rates are low and all patients relapse, due to cellular and soluble immunosuppressive mechanisms. These immunosuppressive mechanisms will be better characterized and their involvement in therapeutic responses in non-small cell lung cancers (NSCLC). Indeed, large transcriptomic analysis of different subsets of immunosuppressive cells will performed, correlating them to clinical outcome in a cohort of stage III disease, treated by radiochemotherapy and immunotherapy as maintenance, and stage IV treated by immunotherapy as first-line treatment. Furthermore, we will analyse cellular mechanisms by in vitro studies, assessing the effect of immunosuppressive cells, provided by fresh tumor samples, on phenotype and functions of lung cancer cell lines. The aim of this study is to better characterize immunosuppressive landscape of NSCLC and mechanisms involved in their protumor functions.

DETAILED DESCRIPTION:
In recent years, immune-based therapies have revolutionized the field of oncology by significantly improving survival of cancer patients. Despite sustained responses, only 20% to 40% of cancer patients respond. It has become clear that the immunosuppressive environment induced by tumor through cellular and/or soluble pathways critically contribute to hinder efficient antitumor immunity. The inhibition of these immunosuppressive networks thus represents an essential prerequisite for the improvement of responses to anticancer immunotherapies. Several immune and non -immune cell populations have been identified as key actors of tumor-induced immunosuppression, among which are myeloid-derived suppressor cells (MDSC), and cancer associated fibroblasts (CAF). However, in non-small cell lung cancers (NSCLC), the phenotypic characteristics and the prognostic role of these cells, the mechanisms underlying their immunosuppressive functions, and their role in dampening the efficacy of immunotherapies in clinical practice are less characterized. The aim of this project is to better characterize these different immunosuppressive subpopulations, and to study their role promoting NSCLC development and resistance to immunotherapies.

First the tumor CAF and immunosuppressive microenvironment using single cell RNA sequencing will be characterized (objective 1a). After identification of phenotypic markers, the immunosuppressive landscape of stage III NSCLC on a lung cancer cohort treated at Bordeaux University Hospital will be analysed, and data on CAF, MDSC and immune infiltration will be correlated with tumor characteristics and cancer outcome (objective 1b). Finally, the pro-tumor functions of CAF isolated from lung cancer patients will be assessed in vitro (objective 2).

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients
* lung carcinoma surgically treated by surgery only (objectives 1a and 2), or stage III lung carcinoma treated by concomitant radiochemotherapy followed by durvalumab (maintenance) treated between September 2018 and december 2021 (objective 1b)

Exclusion Criteria:

* patient receiving chemotherapy, radiotherapy or immunotherapy in the neoadjuvant setting (all objectives)
* patient with previous cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung carcinoma surgically treated by surgery only, or stage III lung carcinoma treated by concomitant radiochemotherapy followed by durvalumab (maintenance) treated between September 2018 and december 2021
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of immune infiltration and phenotypic and functional characteristics of the different cell subgroups isolated from fresh tumors | At the time of surgery only, when fresh tumor is resected
  Exploratory analysis of the immune infiltration (phenotype and function of immunosuppressive and antitumor immune cells) and of the cancer-associated fibroblasts through a transcriptomic analysis of fresh resected lung carcinoma, comparing patients with lymph node involvement or not. Bioinformatics analysis of gene panels

SECONDARY OUTCOMES:
Correlation between the infiltration of CAF and immunosuppressive immune cells and with clinicopathological parameters and patient prognosis (relapse free-survival, overall survival) in stage III NSCLC exposed to immunotherapy | Between September 2018 and December 2021, receiving concomitant radiochemotherapy followed by durvalumab (maintenance)
  Analyze CAF and immunosuppressive immune infiltration in a cohort of unresectable stage III lung carcinoma treated with radiochemotherapy followed by immunotherapy, assessing correlation between immunosuppressive subpopulations and clinical parameters and patient outcome. We will use a multiplexing immunofluorescence assay
Comparative analysis of the modifications of phenotype and functions of MDSC and T lymphocytes when exposed to CAF extracted from patient tumor tissue | At the time of surgery only, when fresh tumor is resected
  Functional in vitro studies of the effect of CAF on phenotype and function of T lymphocytes and of MDSC being extracted from resected NSCLC prospectively collected

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux - Hôpital Saint-André, Service d'Oncologie Médicale, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No